CLINICAL TRIAL: NCT00729040
Title: Enhancing Adherence to an Internet-Mediated Walking Program by Building Online Communities
Brief Title: Enhancing Adherence by Building Online Communities
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Robert Wood Johnson Foundation (Other)
Responsible Party: Caroline Richardson, MD, University of Michigan Health System Dept. of Family Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 57408
Record Dates: First submitted 2008-08-01; First posted 2008-08-06 (Estimated); Last update posted 2009-01-29 (Estimated); Status verified 2009-01

CONDITIONS: Type 2 Diabetes; Coronary Artery Disease; Obesity
Keywords: heart; weight; Overweight; bmi; diabetes; type 2; diabetic; walk; walk*; diab*; obese; exercise; activity; coronary; pedometer
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Coronary Artery Disease; Obesity; Body Weight; Overweight; Diabetes Mellitus; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Stepping Up to Health only
  Interventions: Behavioral: Stepping Up to Health
- 2 (Experimental): Stepping up to Health PLUS online message boards to talk with other participants
  Interventions: Behavioral: Stepping Up to Health

INTERVENTIONS:
Behavioral: Stepping Up to Health — Internet-mediated walking program with pedometers, goal-setting and tailored messaging

SUMMARY:
The purpose of this study is to determine whether online peer support will increase adherence to an internet-based pedometer walking program.

DETAILED DESCRIPTION:
Stepping Up to Health with eCommunities is a study that takes what we already know about motivating sedentary, chronically ill people to walk, and begins to explore what it takes to keep people motivated to exercise over time: the ability to self-monitor behavior with accurate ecological momentary assessments.

We have theorized that peer support, monitoring and competition are ways in which people can stay motivated to meet their walking goals; thus, we have built into this intervention online forums for participants to communicate with each other and garner support, as well as a pilot one-to-many competitive game based on the percent of an individual's goal met.

Our research question is whether online community participation can increase adherence to an Internet-mediated walking program, which consists of an uploading pedometer, and going to a website to receive graphical and textual feedback as to whether participants are meeting gradually increasing walking goals. Three hundred participants will spend four months in this randomized, controlled trial to compare the intervention alone to the intervention plus online community support.

ELIGIBILITY:
Inclusion Criteria:

* Must have one or more of the following: Coronary artery disease (CAD); BMI 25 or higher; Type 2 diabetes
* Must be sedentary, defined by less than 150 minutes of self-reported activity per week
* Must be 18 or older
* Must have access to a computer with an Internet connection, a USB port, and Windows 2000 (latest service pack), XP or Vista
* Must be a regular email user (checking weekly)
* Must be able to communicate in English

Exclusion Criteria:

* Pregnant
* Cannot walk a block (self-report)
* Not competent to sign consent
* Unable to obtain medical clearance from a treating physician (primary care, cardiologist, endocrinologist)
* Type 1 diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2008-01; Primary Completion 2008-10 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
Total steps | last 30 days of intervention

SECONDARY OUTCOMES:
dropout rate | Four months
days and hours pedometer worn | four months
login frequency | four months
upload frequency | four months
content of posts (qualitative) | four months

CONTACTS AND LOCATIONS:
Overall Officials: Caroline R Richardson, MD, Principal Investigator — University of Michigan Health System Dept. of Family Medicine

REFERENCES:
- [Derived] Richardson CR, Buis LR, Janney AW, Goodrich DE, Sen A, Hess ML, Mehari KS, Fortlage LA, Resnick PJ, Zikmund-Fisher BJ, Strecher VJ, Piette JD. An online community improves adherence in an internet-mediated walking program. Part 1: results of a randomized controlled trial. J Med Internet Res. 2010 Dec 17;12(4):e71. doi: 10.2196/jmir.1338. PMID 21169160
- [Derived] Buis LR, Janney AW, Hess ML, Culver SA, Richardson CR. Barriers encountered during enrollment in an internet-mediated randomized controlled trial. Trials. 2009 Aug 23;10:76. doi: 10.1186/1745-6215-10-76. PMID 19698154